CLINICAL TRIAL: NCT05580458
Title: Phase 1/2 Open-label Trial of Safety and Zoster Immunogenicity Evaluation for People With HIV With CD4 Counts Under and Above 300 and Healthy Volunteers Following Shingrix Vaccination (ZEUS)
Brief Title: Safety and Immunogenicity of Recombinant Varicella Zoster Virus Vaccine in People With HIV Who Have a CD4 Count Less Than 300 or Greater Than or Equal to 300 and a Healthy Control Population
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10000866; 000866-I
Record Dates: First submitted 2022-10-08; First posted 2022-10-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12-18

CONDITIONS: Herpes Zoster
Keywords: HERPES ZOSTER; Shingrix Vaccine
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Shingrix (Experimental): Shingrix will be administered in two 0.5-mL doses approximately 2 months apart.
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: Shingrix — Shingrix is a recombinant, adjuvanted vaccine for prevention of herpes zoster. It is supplied as lyophilized recombinant VZV surface gE antigen for reconstitution with AS01B adjuvant suspension. Each Shingrix dose will be 0.5mL and administered by IM injection in the deltoid region of the upper arm.

SUMMARY:
Background:

Shingles is a painful, blistering rash caused by the same virus that causes chickenpox. Shingrix is a vaccine approved to prevent shingles in healthy adults over age 50 and in immunocompromised adults over age 18. Researchers want to learn more about how people with HIV respond to Shingrix.

Objective:

To learn how Shingrix affects the immune response in people with HIV.

Eligibility:

People aged 18 years and older with HIV. Healthy people aged 50 years or older are also needed.

Design:

Participants will have at least 4 clinic visits in 1 year.

Participants will be screened. They will have a physical exam with blood and urine tests.

At their first visit, participants will receive Shingrix as a shot in the upper arm. They will have a rectal swab; a cotton swab will be inserted into the rectum and rotated gently to collect bacteria.

Participants will receive a second shot of Shingrix 2 months after the first one. They will visit the clinic again 3 and 12 months after the first shot.

Participants will receive a 28-day memory tool. They will write down their symptoms between clinic visits. They will have up to 4 phone calls to talk about side effects of the shot.

Participants may undergo apheresis: They will lie still while blood is drawn from a needle in one arm. The blood will pass through a machine that separates out the white blood cells. The remaining blood will be given back through a second needle in their other arm.

DETAILED DESCRIPTION:
Study Description:

This phase 1/2 open-label study will evaluate the safety and immunogenicity of the Shingrix recombinant varicella zoster virus vaccine (RZV) in people with HIV (PWH) aged 18 years and older and healthy volunteers aged 50 years and older. Shingrix will be administered by intramuscular (IM) injection during visits at months 0 and 2, and blood will be collected prior to each dose and at follow-up visits at months 3 and 12. Study evaluations will include assessment of adverse events (AEs) by physical examination, safety laboratory evaluations, and participant memory tool, and assessment of response in research immunogenicity assays on blood.

Objectives:

Primary Objective:

-Assess vaccine immunogenicity after administration of a full Shingrix series schedule in PWH based upon CD4 count < 300 and >= 300.

Secondary Objectives:

* Assess vaccine immunogenicity after administration of a full Shingrix series schedule in PWH by age (< 50 and >= 50 years).
* Compare vaccine immunogenicity in PWH versus healthy volunteers.
* Evaluate grade 3 and 4 safety responses in PWH, based upon CD4 count (< 300 and >= 300), and healthy volunteers.
* Evaluate grade 3 and 4 safety responses in PWH, based upon age (< 50 and >= 50), and healthy volunteers.

Tertiary/Exploratory Objectives:

* Compare immune cell responses in PWH, based upon CD4 count (< 300 and >= 300), and healthy volunteers.
* Compare immune cell responses in PWH, based upon age (< 50 and >= 50 years), and healthy volunteers.
* Assess vaccine immunogenicity by varicella zoster serostatus.
* Assess zoster reactivation.
* Correlate the microbiome profile with vaccine responses.

Endpoints:

Primary Endpoint:

-Fold change of anti-glycoprotein gE (anti-gE) antibody concentrations evaluated regularly through the end of study (months 3 and 12) by CD4 count (< 300 and >= 300) run by GlaxoSmithKline (GSK).

Secondary Endpoints:

* Fold change of anti-gE antibody concentrations evaluated regularly through the end of study (months 3 and 12) by age (< 50 and >= 50) run by GSK.
* Fold change of anti-gE antibody concentrations evaluated regularly through the end of study (months 3 and 12) in PWH and healthy volunteers run by GSK.
* Grade 3 and/or Grade 4 Shingrix AEs (solicited and unsolicited local and systemic).

Tertiary/Exploratory Endpoints:

* T-cell assays and phenotypes evaluated regularly through end of study.
* Varicella zoster serostatus as determined by IgG and IgM antibody levels.
* Number of episodes and severity of zoster reactivation (including extradermatomal complications such as neurologic or ophthalmologic complications and adverse sequelae such as post herpetic neuralgia).
* Baseline microbiome profile.

ELIGIBILITY:
* INCLUSION CRITERIA:

General Inclusion Criteria:

Individuals must meet all of the following criteria to be eligible for study participation:

* Able to provide informed consent.
* Participants of childbearing potential must agree to use at least 1 acceptable method of contraception when engaging in sexual activities that can result in pregnancy, beginning at screening through month 3. Acceptable methods of contraception include the following:

  * Hormonal contraception.
  * Male or female condom.
  * Diaphragm or cervical cap with a spermicide.
  * Intrauterine device.
* Has a primary care provider.

Additional Inclusion Criteria for People with HIV:

* PWH must also meet all the following criteria to be eligible for study participation:
* >= 18 years of age.
* Seropositive for HIV-1 (documented or confirmed at screening).
* Documented viral load < 100 copies/mL within 30 days of screening and documented suppression < 40 copies/mL within 6 months of screening.
* Currently on a stable antiretroviral regimen (minimum of 6 months of a stable ART regimen; changes for side effects, drug interaction, or convenience allowed), or is an elite controller (maintains undetectable viral loads in the absence of any treatment for a period of one year prior to screening visit).
* No active/uncontrolled opportunistic infections (patients on chronic maintenance therapy would be considered as controlled).

Additional Inclusion Criteria for Healthy Volunteers:

Healthy volunteers must also meet all of the following criteria to be eligible for study participation:

* >= 50 years of age.
* No uncontrolled chronic medical issues that per the discretion of the PI or designee would compromise the safety of the research participant.
* No underlying immunodeficiencies (including negative HIV test at screening).

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

* Previous receipt of Shingrix vaccine at any time.
* Receipt of Zostavax within the past 12 months.
* History of severe allergic reaction to any component of Shingrix.
* Diagnosed varicella or herpes zoster episode within the past 1 month. Subject will be eligible for SHINGRIX vaccine once symptoms of herpes zoster episode have resolved.
* Immunocompromised (other than HIV for the PWH cohort) within the past 6 months (eg, due to a malignancy other than skin cancer).
* Current moderate or severe acute illness (ie, febrile illness, seizure, myocardial infarction, cerebrovascular accident, pulmonary embolism) that in the opinion of the principal investigator, would make the subject unsuitable for the study.
* Pregnancy or breastfeeding.
* Receipt of an investigational agent, investigational vaccine, or licensed live virus vaccine within 30 days prior to screening.
* Planned receipt of any vaccine (investigational or ACIP-recommended) between months 0 and 2 except for the tetanus, diphtheria, and pertussis vaccine [TDaP], Pneumovax, inactivated influenza vaccines, and COVID-19 vaccine which may be given at least 8 days before and/or at least 14 days after each study agent injection (at month 0/month 2).
* Administration of immunoglobulins or any blood products within 90 days preceding the first dose of vaccine or planned administration during the study period.
* Chronic administration (>= 15 consecutive days) of immunosuppressive or other immune-modifying drugs within 6 months before screening. (Prednisone < 20 mg/day or equivalent, corticosteroid nasal spray or inhaler, and topical steroids are not exclusionary).
* Uncontrolled psychiatric disease per physician evaluation, current substance use, or inappropriate conduct unsuitable for a research study.
* Any condition that could compromise, in the investigator's opinion, the participant's safety or the study outcomes.

Participants will be selected in an equitable manner from the available pool of potentially eligible individuals, without regard to factors such as sex, race, ethnicity, socioeconomic status, etc, except for age.

Medical record review may be used for determining eligibility. If a clinical laboratory evaluation is available for review at the screening timepoint, but was obtained prior to protocol consent, the laboratory test does not have to be repeated for the purposes of confirming eligibility under the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Fold change of anti-gE antibody concentrations evaluated regularly through the end of study (months 3 and 12) by CD4 count (< 300 and >= 300) | Months 3 and 12
  Assess vaccine immunogenicity after administration of a full Shingrix series schedule in PWH based upon CD4 count < 300 and >= 300.

SECONDARY OUTCOMES:
Fold change of anti-gE antibody concentrations evaluated regularly through the end of study in PWH and healthy volunteers | Months 3 and 12
  Compare vaccine immunogenicity in PWH versus healthy volunteers.
Grade 3 and/or Grade 4 Shingrix ARs (solicited and unsolicited local and systemic). | Through the end of the study
  Evaluate grade 3 and 4 safety responses in PWH, based upon age (< 50 and >= 50), and healthy volunteers.
Grade 3 and/or Grade 4 Shingrix ARs (solicited and unsolicited local and systemic). | Through the end of the study
  Evaluate grade 3 and 4 safety responses in PWH, based upon CD4 count (< 300 and >= 300), and healthy volunteers.
Fold change of anti-gE antibody concentrations evaluated regularly through the end of study by age (< 50 and >= 50) | Months 3 and 12
  Assess vaccine immunogenicity after administration of a full Shingrix series schedule in PWH by age (< 50 and >= 50 years).

CONTACTS AND LOCATIONS:
Overall Officials: Maura M Manion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lal H, Cunningham AL, Godeaux O, Chlibek R, Diez-Domingo J, Hwang SJ, Levin MJ, McElhaney JE, Poder A, Puig-Barbera J, Vesikari T, Watanabe D, Weckx L, Zahaf T, Heineman TC; ZOE-50 Study Group. Efficacy of an adjuvanted herpes zoster subunit vaccine in older adults. N Engl J Med. 2015 May 28;372(22):2087-96. doi: 10.1056/NEJMoa1501184. Epub 2015 Apr 28. PMID 25916341
- [Background] Berkowitz EM, Moyle G, Stellbrink HJ, Schurmann D, Kegg S, Stoll M, El Idrissi M, Oostvogels L, Heineman TC; Zoster-015 HZ/su Study Group. Safety and immunogenicity of an adjuvanted herpes zoster subunit candidate vaccine in HIV-infected adults: a phase 1/2a randomized, placebo-controlled study. J Infect Dis. 2015 Apr 15;211(8):1279-87. doi: 10.1093/infdis/jiu606. Epub 2014 Nov 3. PMID 25371534
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000866-I.html